CLINICAL TRIAL: NCT06023212
Title: Tranexamic Acid Use for Bleeding Prevention in the Surgical Treatment of Metastatic Spinal Tumor in Lung Cancer Patients: a Triple Blinded, Randomized Controlled Trial to Assess the Efficacy of Tranexamic Acid for Hemostasis
Brief Title: Tranexamic Acid Use for Bleeding Prevention in the Surgical Treatment of Metastatic Spinal Tumor in Lung Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022_LHY
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Metastasis Spinal Tumor
Keywords: Tranexamic Acid; blood loss; seperation surgery
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tranexamic acid group (Experimental): injection of 2 bottles of tranexamic acid (1g/bottle) before making incision; tranexamic acid soaked gauze applied to the wound before closing the wound; Intravenous injection of tranexamic acid 3 times (every 8 hours）within 24 hours after operation；
  Interventions: Drug: Tranexamic Acid
- SPSS group (Placebo Comparator): injection of 2 bottles of stroke-physiological saline solution（SPSS）before making incision; SPSS soaked gauze applied to the wound before closing the wound; Intravenous injection of SPSS 3 times (every 8 hours）within 24 hours after operation；
  Interventions: Drug: stroke-physiological saline solution (SPSS)

INTERVENTIONS:
Drug: Tranexamic Acid — IV drip of 2 bottles of tranexamic acid (2g) before making incision during surgery；
  1g tranexamic acid soaked gauze applied to the wound for 5 minintes before suture； patients were administered IV drip of tranexamic acid 3 times (every 8 hours)within 24 hours after surgery.
  Arms: tranexamic acid group
Drug: stroke-physiological saline solution (SPSS) — IV drip of 2 bottles of saline before making incision during surgery； saline soaked gauze applied to the wound for 5 minintes before suture； patients were administered IV drip of saline 3 times (every 8 hours)within 24 hours after surgery.
  Arms: SPSS group

SUMMARY:
Massive blood loss occurs in metastatic spinal tumor resection and may cause severe complications. The objective of this study is to investigate whether the use of tranexamic acid will reduce perioperative and postoperative bleeding when compared to those without use of tranexamic acid.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as metastatic carcinoma of the thoracolumbar spine
* solitary neoplasm involve only one segment of spine
* patients underwent separation surgery

Exclusion Criteria:

* coagulation function was abnormal preoperatively
* patients are allergic to tranexamic acid
* neoplasm involve more than one segment of spine
* patients with rich blood supply who need embolization

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
total blood loss | measured 3 days postoperatively
  the loss of total blood volume caused by various operations (mainly during surgical operations) throughout the entire treatment process.
  Total blood volume = preoperative blood volume *（preoperative hematocrit - hematocrit 3 days postoperatively）
Intraoperative blood loss | 1 day (measured once after surgery)
  Refers to the total blood loss of a patient experienced during operation from skin incision to wound suture.
  Intraoperative blood loss = intraoperative drainage volume - intraoperative flushing volume + blood loss estimation using gauze (calculated as 10 cm × 10 cm gauze absorbs 10 ml)

SECONDARY OUTCOMES:
allogeneic transfusion blood volume | 1 day (measured once during surgery)
  amount of allogeneic transfusion blood volume needed during operation

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided